CLINICAL TRIAL: NCT02293122
Title: To Investigate Agreement Between the EM-3000 and the Predicate Device NonCon Robo Pachy (F&A) (CellChek XL).
Status: Completed | Type: Observational
Sponsor: Tomey Corporation (Industry)
Collaborators: Ohio State University (Other); R. P. Chiacchierini Consulting, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 602-a01
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Observational group exposure to three test devices and one comparative device. The test Konan Non-con Robo Pachy F&A Specular Microscope.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Intervention is observational to two different diagnostic devices for which comparative readings of the corneal endothelium are being measured; the test device- the EM-3000 Specular Microscope against the Konan Robo-pachy F&A Specular Microscope.

SUMMARY:
The purpose of this study is to evaluate the precision and agreement of the study device, a specular microscope, in comparison to a currently commercially available specular microscope in establishing substantial equivalence of the two devices in clinical use for diagnostic purposes of the human cornea.

DETAILED DESCRIPTION:
The observational clinical investigation is intended to measure agreement between two diagnostic instruments of the eye's corneal endothelium. The study device is the EM-3000 specular microscope and the control device is the NonCon Robo Pachy (F&A) (CellChek XL) specular microscope. Both instruments measure corneal endothelial cell layer parameters including cell density, coefficient of variation, percent hexagonality, and central thickness.

The primary variable is the measurement of agreement between the two instruments for the four parameters described. The secondary variables include repeatability (intra-investigator) and reproducibility both inter-investigator, and inter-instrument.

Additionally, measurements of agreement will be made on the EM-3000 using automated analysis with and without touch-up.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with one of the following corneal conditions:

Non-pathologic younger eyes (18-50 yrs) Non-pathologic older eyes (51-80 yrs) Pathologic adult eyes (29-80)

Exclusion Criteria

1. Seriously ill or unconscious subject, mentally ill person, mentally handicapped person, person who is unable to read or write.

   * Non-Pathologic subjects who have the following conditions :
2. History of corneal transplant
3. Long term Fuch's dystrophy (and other corneal endothelial dystrophy)
4. Guttata
5. History of cataract or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device
6. Long term PMMA contact lens use longer than 5 years

   -Pathologic subjects
7. Keratoconus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study plan calls for 75 subjects divided into three sub-groups, young healthy (18-50 yrs), older healthy (51-80 yrs), and pathologic adults (29-80 years).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Agreement Between EM-3000 and NonCon Robo Pachy F&A (CellChek XL) | 1 day visit per subject.
  For Agreement between the two instruments, outcome measures include endothelial cell density (/mm2), coefficient of variation between the two instruments (SD x CD x 10-6, and percent hexagonality of cells in the measured visible field of view between the two instruments.

SECONDARY OUTCOMES:
Investigate Repeatability and Reproducibility between the EM-3000 and NonCon Robo Pachy F&A (CellChek XL) Specular Microscopes | 1 day visit per subject.
  To investigate repeatability (intra-investigator) in the EM-3000 specular microscope in the four outcome measures of the corneal endothelium as well as corneal thickness.
  To investigate reproducibility (inter-investigator/instrument) of the EM-3000 specular microscope in the four outcome measures of the corneal endothelium and corneal thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bailey, OD, Principal Investigator — Professor, College of Optometry
Locations (1):
- Ohio State University, Columbus, Ohio, United States